CLINICAL TRIAL: NCT00218049
Title: Phase 1, Double-blind, Placebo-controlled Assessment of Interactions Between 2 Doses of Cocaine and Three Doses of Escalating Vanoxerine (GBR 12909) in Cocaine Using Volunteers
Brief Title: Interaction Between Vanoxerine (GBR 12909) and Cocaine in Cocaine Dependent Individuals
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issue of priority of resources
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Responsible Party: F. Gerard Moeller, M.D., University of Texas Medical School at Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-09262-10; P50-09262-10; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Cocaine Abuse; Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — vanoxerine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 50 mg of GBR 12909
  Interventions: Drug: GBR 12909
- 2 (Experimental): 75 mg of GBR 12909
  Interventions: Drug: GBR 12909
- 3 (Experimental): 100 mg of GBR 12909
  Interventions: Drug: GBR 12909

INTERVENTIONS:
Drug: GBR 12909 — 50mg GBR 12909 over 12 days
  Arms: 1
Drug: GBR 12909 — GBR 12909 75 mg over 12 day period
  Arms: 2
Drug: GBR 12909 — GBR 12909 100 mg over 12 day period
  Arms: 3

SUMMARY:
Cocaine dependence is a major public health problem; an effective primary treatment for cocaine dependent individuals has yet to be found. The purpose of this study is to determine the safety and effects of vanoxerine (GBR 12909) in treating cocaine dependent individuals.

DETAILED DESCRIPTION:
Cocaine is a strong central nervous system stimulant that is widely abused throughout the United Sates. Due to its widespread use, it is important to develop an effective treatment for cocaine dependence. Dopamine transporters (DAT) play an important role in the addictive nature of cocaine; the use of compounds that target DAT may be effective in treating cocaine dependent individuals. Research shows that GBR 12909 has a strong affinity for DAT. The purpose of this study is to determine the safety and potential interaction of GBR 12909 and cocaine in cocaine dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine dependence
* Not currently seeking treatment for cocaine dependence
* Currently uses cocaine, as determined by a self-report and a positive urine test for cocaine, within 30 days prior to study entry
* Within 20 % of ideal body weight, and weighs at least 100 lbs
* Good general health
* Normal electrocardiogram
* Willing to use acceptable methods of contraception for the duration of the study

Exclusion Criteria:

* Current or history of a major psychiatric illness, other than drug dependence or disorders secondary to drug abuse
* Meets DSM-IV criteria for dependence on any drugs other than cocaine, marijuana, nicotine, or alcohol
* Physiologically dependent on alcohol and requires medical detoxification
* Use of prescription drugs within 14 days prior to study entry
* Use of non-prescription drugs within 7 days prior to study entry
* If female, used an oral contraceptive, Depo-Provera, Norplant, or intrauterine progesterone contraceptive system, within 30 days prior to study entry
* Pregnant or breastfeeding
* History of liver disease
* Current elevated aspartate aminotransferase or alanine aminotransferase levels
* Donated a unit of blood within 4 weeks prior to study entry
* Participated in any other clinical investigation within 4 weeks prior to study entry
* History of any illness or behavior that, in the opinion of the investigator, might interfere with the study
* Family history of early significant cardiovascular disease
* Exhibits Hepatitis B surface antigen or Hepatitis C antibody
* HIV infected
* Syphilis
* Active tuberculosis
* Adult asthma
* Chronic obstructive pulmonary disease
* Unable to distinguish between 20 mg and 40 mg of intravenous cocaine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Medication effects, including frequency of adverse events | 12 days of trial

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States